CLINICAL TRIAL: NCT02136095
Title: Promising Initial Experience With Intra-operative Fluorescent Cholangiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Søren S. Larsen, MD, PhD, Hvidovre University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IFC_Feasibility_study
Record Dates: First submitted 2014-05-07; First posted 2014-05-12 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Gall Stone Disease
Keywords: Fluorescent cholangiography; Laparoscopic cholecystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IFC-group (Experimental): The investigators included patients undergoing laparoscopic cholecystectomy by a single surgeon between September and December 2013 at a single centre university department with unrestricted referral of patients. The included patients represented all patients undergoing laparoscopic cholecystectomy by one surgeon during the study period. All patients underwent intra-operative fluorescent cholangiography (IFC) with concomitant angiography, according to a standardized protocol, during their laparoscopic cholecystectomy.
  Interventions: Procedure: Intraoperative fluorescent cholangiography (IFC)

INTERVENTIONS:
Procedure: Intraoperative fluorescent cholangiography (IFC) — A standardized protocol with IFC including concomitant angiography was performed during laparoscopic cholecystectomy.

SUMMARY:
Intraoperative fluorescent cholangiography (IFC) with concomitant fluorescent angiography is a recently developed method for non-invasive visualisation of the relevant anatomy during laparoscopic cholecystectomy. The objective of this study was to assess the time required by routine-use of IFC and to evaluate success-rate of the procedures.

Methods Thirty-five patients scheduled for laparoscopic cholecystectomy and operated by the same surgeon were consecutively enrolled. A standardized protocol with IFC including concomitant angiography was performed during laparoscopic cholecystectomy. Intra-operative time-registration and exposure of predefined anatomical structures were recorded.

ELIGIBILITY:
Inclusion criteria:

* Age > 18 years
* Scheduled for acute- or elective laparoscopic cholecystectomy
* Informed consent

Exclusion criteria:

* Known iodine-hypersensitivity
* Liver- or renal insufficiency
* Known thyrotoxicosis
* Pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Time expenditure of IFC with concomitant angiography. | Four months
  Intra-operative fluorescent-imaging-mode-time was registered by a study-nurse during the operations (performed between september and december 2013)

SECONDARY OUTCOMES:
Success-rate of the IFC-procedures. | Four months
  The operating surgeon completed a structured questionnaire immediately after each operation regarding anatomical identification by IFC (visible cystic duct, -common bile duct, -common hepatic duct, -right and left hepatic ducts, -cystic artery, -aberrant bile ducts, and/or other abnormalities).
  Successful IFC was defined as exposure of the junction between the cystic duct, common bile duct and common hepatic duct by IFC. Success-full fluorescent angiography was defined as adequate visualisation of the cystic artery within Calot´s triangle by the method.

CONTACTS AND LOCATIONS:
Overall Officials: Søren Larsen, MD, PhD, Principal Investigator — Gastroenheden, Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Hvidovre, Denmark

REFERENCES:
- [Derived] Larsen SS, Schulze S, Bisgaard T. Non-radiographic intraoperative fluorescent cholangiography is feasible. Dan Med J. 2014 Aug;61(8):A4891. PMID 25162446